CLINICAL TRIAL: NCT02847000
Title: p53/p16-Independent Epigenetic Therapy With Oral Decitabine/Tetrahydrouridine for Advanced Pancreatic Cancer That Has Progressed Through One or More Lines of Therapy
Brief Title: p53/p16-Independent Epigenetic Therapy With Oral Decitabine/Tetrahydrouridine for Pancreatic Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yogen Saunthararajah (Other)
Responsible Party: Sponsor-Investigator, Yogen Saunthararajah, Professor, Hematology and Oncology, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2216
Record Dates: First submitted 2016-07-25; First posted 2016-07-27 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
Keywords: Decitabine; Tetrahydrouridine; Epigenetic Therapy
MeSH Terms: interventions — Tetrahydrouridine; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Decitabine + Tetrahydrouridine (Experimental): Tetrahydrouridine (THU) is supplied as 250 mg/capsule, Decitabine (Dec) as 5 mg/capsule.
  Interventions: Drug: Tetrahydrouridine; Drug: Decitabine

INTERVENTIONS:
Drug: Tetrahydrouridine — Starting dose is by weight:
  THU is supplied as 250 mg/capsule Weight 40-60kg = 2 capsules of Tetrahydrouridine. Weight 61-80kg = 3 capsules of THU. Weight 81-100kg or higher = 4 capsules of THU.
  Timing between THU and Dec, Frequency of administration: Oral THU capsules followed 60 minutes later by oral Dec capsules are ingested 2X/week on consecutive days. Treatment on protocol monitoring continues for 52 weeks, however, subjects will have the option to continue beyond this period if it judged to be in their interests.
  Other Names: THU
Drug: Decitabine — Starting dose is by weight:
  DEC is supplied as 5 mg/capsule. Weight 40-60kg = 2 capsules of Decitabine. DEC capsules are ingested ~60 minutes after THU capsules. Weight 61-80kg = 3 capsules of DEC. DEC capsules are ingested ~60 minutes after THU capsules. Weight 81-100kg or higher = 4 capsules of DEC. DEC capsules are ingested ~60 minutes after THU capsules.
  Timing between THU and Dec, Frequency of administration: Oral THU capsules followed 60 minutes later by oral Dec capsules are ingested 2X/week on consecutive days. Treatment on protocol monitoring continues for 52 weeks, however, subjects will have the option to continue beyond this period if it judged to be in their interests.
  Other Names: DEC

SUMMARY:
Patients with pancreatic cancer which has stopped responding to one or more chemotherapy drugs are asked to take part in this study. The study hopes to find out whether decitabine, the drug being studied, will have an effect on pancreatic cancer. The decitabine is being given at a lower dose than its approved use. It is also being given with another drug, tetrahydrouridine (THU), to improve the exposure of your pancreatic cancer cells to decitabine.

The purpose of this study is to determine if the drug combination of decitabine and tetrahydrouridine can recognize a certain DNA target in your cancer. All cells have DNA within them, and tumor cells have abnormal DNA.

DETAILED DESCRIPTION:
Primary Objective The primary goal of this pilot study is to detect decitabine therapy induced DNMT1 protein level decreases with an effect size of 1 using a paired t-test and alpha=0.05. The effect size is defined as the difference in mean DNMT1-protein levels between post-treatment and pre-treatment divided by the standard deviation and is thus a metric of change in the natural units of the distribution, its standard deviation. Our goal is thus to detect drops in DNMT1 of at least one standard deviation.

Secondary Objectives Secondary goals include correlating DNMT1 decreases with clinical response (measured by Response Evaluation Criteria in Solid Tumors [RECIST1.1]), using logistic regression; time to relapse, using a Cox model; tolerability and safety assessment by toxicity characterization using CTCAEv4.

Study Design Single-arm, open-label, proof-of-concept clinical trial in patients with metastatic pancreatic cancer that has progressed on one or more lines of systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven pancreatic carcinoma or adenocarcinoma. Histologies other than carcinoma/adenocarcinoma will not be eligible.
* Subjects must have received one or more prior systemic therapies for this disease, with disease progression or intolerable toxicity precluding further therapy with prior regimen(s).
* Measurable disease per RECIST 1.1.
* ECOG performance status 0 - 2
* Adequate organ function as defined by the following criteria:

  * Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 x laboratory upper limit of normal (ULN)
  * Total serum bilirubin ≤ 2.0 x ULN
  * Absolute neutrophil count (ANC) ≥ 1500/uL
  * Platelets ≥ 75,000/uL
  * Hemoglobin ≥ 8.0 g/dL
  * Serum calcium ≤ 12.0 mg/dL
  * Serum creatinine ≤ 2.9 mg/dL
* Eligible and agreeable for percutaneous biopsy of a primary or metastatic lesion prior to treatment and after approximately 16 weeks of treatment
* Patients with history of brain metastases can be enrolled at a minimum of 2 weeks following the completion of surgery, gamma knife or whole brain radiotherapy. Repeat brain MRI not required for eligibility.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.
* At least two-weeks since receipt of prior standard or investigational therapy.

Exclusion Criteria:

* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, severe peripheral vascular disease (claudication) or procedure on peripheral vasculature, coronary/peripheral artery bypass graft, New York Heart Association grade II or greater congestive heart failure, cerebrovascular accident or transient ischemic attack, clinically significant bleeding or pulmonary embolism.
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness (HIV-positive subjects on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with oral THU-Dec. Appropriate studies will be undertaken in subjects receiving combination antiretroviral therapy when indicated.
* Pregnancy or breastfeeding (pregnant or breastfeeding women are excluded from this study because oral THU-Dec has the potential for teratogenic or abortifacient effects. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with oral THU-Dec, breastfeeding should be discontinued if the mother is treated with oral THU-Dec.
* Other severe acute or chronic medical or psychiatric conditions or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.
* Receiving other investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
DNMT1 protein level decreases with an effect size of 1 | up to 12 months
  Differences will be calculated using a paired t-test and alpha=0.05. The effect size is defined as the difference in mean DNMT1-protein levels between post-treatment and pre-treatment divided by the standard deviation and is thus a metric of change in the natural units of the distribution, its standard deviation. Our goal is thus to detect drops in DNMT1 of at least one standard deviation.

SECONDARY OUTCOMES:
Clinical Response as measured by RECIST 1.1 guidelines | up to 12 months
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Best Overall Response | up to 12 months
  The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria.
Duration of Response | up to 12 months
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started) The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that progressive disease is objectively documented.
Duration of stable disease | up to 12 months
  Stable disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started, including the baseline measurements.
Overall Survival | up to 12 months
  Overall Survival will be calculated as time in days from enrollment (signing of the informed consent) to death.
Progression-Free Survival | up to 12 months
  Progression-free Survival will be calculated as time in days from enrollment (signing of the informed consent) to the earlier of:
  * Death, or
  * Disease progression, by clinical or imaging parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Devendra P Sohal, MD, MPH, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio